CLINICAL TRIAL: NCT02104570
Title: Effects of Muscle Fatigue and Kinesio Taping on Shoulder Joint Position Sense
Brief Title: Effects of Muscle Fatigue and Kinesio Taping on Shoulder Position Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 09102013.011
Record Dates: First submitted 2014-03-24; First posted 2014-04-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fatigue; Proprioception
Keywords: Fatigue; Proprioception; Shoulder
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Control (Other): In this session, participants will be evaluated before and after a muscle fatigue protocol, with no intervention.
  Interventions: Other: Fatigue protocol
- Kinesio taping with tension (Experimental): A kinesio taping technique for the deltoid muscle will be applied before fatigue protocol and removed after in the end of the evaluation session. Subjects will be evaluated before taping, after taping and after the fatigue protocol.
  Interventions: Other: Kinesio taping with tension; Other: Fatigue protocol
- Kinesio taping without tension (Sham Comparator): A kinesio taping technique will be applied on the deltoid muscle without tension (tension is considered to be the therapeutic effect) before fatigue protocol and removed after in the end of the evaluation session. Subjects will be evaluated before taping, after taping and after the fatigue protocol.
  Interventions: Other: Kinesio taping without tension; Other: Fatigue protocol

INTERVENTIONS:
Other: Kinesio taping with tension
  Arms: Kinesio taping with tension
Other: Kinesio taping without tension
  Arms: Kinesio taping without tension
Other: Fatigue protocol

SUMMARY:
The purpose of this study is to investigate the effects of Kinesio Taping on the position sense of shoulder after muscle fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* prior shoulder surgery
* shoulder injury that required rehabilitation in the last 2 years
* shoulder dislocation
* ligamentous laxity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in joint repositioning angle errors | Baseline (in the beginning of the session, without taping), 5 minutes after taping (or equivalent time resting, in the control session) and average of 3 minutes after fatigue protocol.
  The joint repositioning errors will be measured during active repositioning trials of shoulder abduction in scapular plane using an iPod app.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Karduna, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States